CLINICAL TRIAL: NCT05270759
Title: Non-invasive Assessment to Predict Tolerance to Fluid Removal on Intermittent Kidney Replacement Therapy
Acronym: TECHNO-HDF
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: The Kidney Foundation of Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-10134, 21.233
Record Dates: First submitted 2022-02-26; First posted 2022-03-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Kidney Injury; Chronic Kidney Disease Stage 5 on Dialysis; Chronic Kidney Failure; Intradialytic Hypotension; Fluid Overload
Keywords: Relative blood volume monitoring; Hemodialysis; Hemodiafiltration; Venous Doppler
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Hospitalized patients receiving hemodialysis/hemodialfiltration: Adult patients hospitalized in the intensive care unit (ICU) or general ward receiving hemodiafiltration or hemodiafiltration treatments as least 3 times per week with ≥1L of fluid removal per session
  Exclusion criteria:
  * Planned hospital discharge, death, or transition to comfort care within 48 hours according to the attending physician
  * End of active care (awaiting hospital discharge)
  Interventions: Diagnostic Test: Estimated absolute blood volume; Diagnostic Test: Modified VExUS evaluation

INTERVENTIONS:
Diagnostic Test: Estimated absolute blood volume — Baseline absolute blood volume will be inferred based on the change in relative blood volume (RBV) after a single 240mL replacement fluid infusion and then monitored throughout the session via the RBV value.
Diagnostic Test: Modified VExUS evaluation — The presence of at least 2/3 abnormal venous Doppler waveforms at the following sites: Portal vein, hepatic vein, and femoral vein.

SUMMARY:
This prospective cohort study aim to investigate the ability of multiple types of assessments including 1) the modified Venous Excess Ultrasound (VExUS) assessment, 2) non-invasive estimation of absolute blood volume (ABV), and 3) change in carotid Doppler at the start of IKRT to predict IDHE in acutely ill hospitalized patients. The secondary aim will be to determine whether each modality improves the prediction of IHDE compared to the evaluation of the attending physician and whether they also predict cerebral hypoxia during IKRT measured by near-infrared spectroscopy (NIRS). Finally, detailed hemodynamic data including relative blood volume monitoring, tissue oximetry, and other parameters will be collected continuously during IKRT sessions enabling exploratory analyses aimed at identifying hemodynamic phenotypes related to IDHE during IKRT.

DETAILED DESCRIPTION:
Background:

Fluid accumulation and intra-dialytic hypotensive events (IDHE) are independently associated with worse prognosis in patients undergoing intermittent kidney replacement therapy (IKRT), both in the setting of acute kidney injury (AKI) and in patients with end-stage kidney disease (ESKD). An optimal IKRT prescription needs to achieve adequate fluid homeostasis while mitigating the risk of IDHE. However, predicting tolerance to fluid removal is challenging, particularly in acutely ill hospitalized patients in whom intravascular volume and compensatory mechanisms are affected by the presence of acute illness.

The following modalities will be investigated in this study to determine if they predict IDHE during hemodialysis in hospitalized patients:

* The modified VExUS assessment before the hemodialysis session
* Estimation of absolute blood volume during the hemodialysis session
* Removed in protocol version 2.0: Change in carotid Doppler parameters in response to fluid administration at the start of hemodialysis

Objectives:

Primary objective:

To determine whether the studied modalities accurately predicts intradialytic hypotension events (IDHE) in hospitalized patients, including critically ill and non-critically ill patients

Secondary objectives:

To determine whether the studied modalities predict cerebral desaturations events measured by near infra-red tissue oximetry (NIRS) during IKRT To determine if adding information from the studied modalities result in significant improvement in the risk prediction of IDHE when added to the subjective assessment of the attending clinician

Study design:

A cohort of hospitalized patients undergoing hemodiafiltration with ultrafiltration will be monitored during two separate dialysis sessions. The following markers will assessed:

1. Absolute blood volume, estimated based on the change in relative blood volume measured by the Fresenius BVM after infusion of a replacement fluid bolus of 240 mL given 15 minutes after dialysis initiation using the Kron et al method.
2. The modified VExUS from the Doppler assessment of the portal, hepatic, femoral, and splenic vein before the hemodialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient ≥18 year-old
2. Hospitalized at the CHUM in the intensive care unit (ICU) or general ward
3. Receiving or planned ≥3x/week IKRT treatments
4. Planned on-line hemodiafiltration (HDF) or hemodialysis (HD) sessions with ≥1L of fluid removal per session

Exclusion Criteria:

1. Planned hospital discharge, death, or transition to comfort care within 48 hours according to the attending physician
2. End of active care (awaiting hospital discharge)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adults with acute kidney injury or chronic kidney disease requiring hemodialysis with on-line hemodiafiltration.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Intradialytic hypotensive event in the peri-dialytic or post-dialytic period | From the initiation of dialysis to 15 minutes after dialysis
  Intradialytic hypotension will be defined as a drop in systolic blood pressure below 90 mmHg which requires an intervention (dialysis interruption, vasopressor initiation or dosage increase, fluid bolus, interruption of net ultrafiltration, change in body position with therapeutic intent) In patients with a baseline below 90 mmHg, it will be defined as a decrease of more than 10 mmHg from baseline systolic blood pressure.

SECONDARY OUTCOMES:
Intradialytic cerebral desaturation events | From the initiation of dialysis to 15 minutes after dialysis
  >15% decrease in cerebral oximetry (NIRS) measurements relative to baseline value.
Rate of intradialytic hypotension | From enrolment to 14 days
  The proportion of sessions with at least one episode of intradialytic hypotension (as previously defined) within 14 days from enrollment
Mortality rate | From enrolment to 90 days
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: William Beaubien-Souligny, MD PhD, Principal Investigator — CR CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Will require data sharing agreement